CLINICAL TRIAL: NCT01605123
Title: Leipzig Artherobesity Childhood Cohort
Brief Title: Longitudinal Assessment of Cardiovascular and Metabolic Parameters in Obese and Lean Children
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Antje Koerner, Prof. Dr. med., Prof. Dr. med., University of Leipzig
Other Study IDs: KFO152/SFB1052-C5
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Obesity
Keywords: endothelial function; children; obesity; cardiovascular dysfunction; carotid intima media thickness; blood pressure; oral glucose tolerance test
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples, samples from oral glucose tolerance tests (oGTT), EDTA/DNA samples, primary cells (endothelial progenitor cells), peripheral blood mononuclear cells), urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lean children: n=100 (anticipated), n=70 currently Age: 6-25 years BMI-SDS: -1.88 to +1.23 , currently -0.25±0.77; Height-SDS: > - 2 SDS, currently 0.03±1.07;
- Obese children: n=106 Age: 6-25 years BMI-SDS: >1.23 , currently 2.41±0.52; Height-SDS: > - 2 SDS, currently 0.80±1.18;
- Obese Exercise Group: Obese children will engage in increased physical activity (one to two lessons per week) at 40-60 and 60-80% of maximal exercise capacity (n=50 each anticipated). Within the frame of the study we will assess the effect of the exercise on cardiovascular outcomes.
- Classical Lifestyle Intervention: Obese children will receive a classical lifestyle intervention, including dietary, activity and psychosocial counselling (n=50 anticipated). Within the frame of the study we will assess the effect of the exercise on cardiovascular outcomes.

SUMMARY:
The investigators hypothesize that cardiovascular and metabolic alterations due to obesity already manifest at childhood age.

To identify these alterations and risk factors, the investigators have established a cohort of 177 healthy obese and lean control children, age ranging from 6y to 18y, for evaluation of cardiovascular and metabolic parameters, as well as quantification of biomarkers of obesity and inflammation. Follow-up analyses are planned after 2 years (completed) and additionally after 5, 7 and 9 years.

In addition, the investigators will assess the effects of increased physical activity and exercise on cardiovascular function.

ELIGIBILITY:
Inclusion Criteria:

* height -2 to +2 SDS
* pubertal stage adequate for age
* no medications
* written consent of guardians and children≥12y
* weight ≥ -2 SDS

Exclusion Criteria:

* secondary/syndromal obesity
* known existing hypertension
* chronic disease (eg. errors of metabolism)
* acute illness (eg. respiratory tract infection)
* previous hypertensive or antidiabetic treatment- weight loss attempts 6 weeks prior to assessment

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obese children from our out-patient department in Leipzig, Germany Lean children community-based from Leipzig
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
cardiovascular dysfunction | 7 years
  Assessment of endothelial function, carotid intima media thickness, blood pressure, echocardiography, exercise capacity, insulin sensitivity by oGTT, serum lipids

CONTACTS AND LOCATIONS:
Overall Officials: Antje Körner, MD, Principal Investigator — University of Leipzig
Locations (2):
- Germany (2):
  - LIFE Leipzig Research Centre for Civilization Diseases, University of Leipzig, Leipzig, Saxony
  - University Leipzig Medical Center, Department of Women and Child Health, Center for Pediatric Research, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korner A, Kratzsch J, Gausche R, Schaab M, Erbs S, Kiess W. New predictors of the metabolic syndrome in children--role of adipocytokines. Pediatr Res. 2007 Jun;61(6):640-5. doi: 10.1203/01.pdr.0000262638.48304.ef. PMID 17426657
- [Result] Landgraf K, Friebe D, Ullrich T, Kratzsch J, Dittrich K, Herberth G, Adams V, Kiess W, Erbs S, Korner A. Chemerin as a mediator between obesity and vascular inflammation in children. J Clin Endocrinol Metab. 2012 Apr;97(4):E556-64. doi: 10.1210/jc.2011-2937. Epub 2012 Mar 21. PMID 22438234
- [Result] Raschpichler MC, Sorge I, Hirsch W, Mende M, Sergeyev E, Kruber D, Koerner A, Schick F. Evaluating childhood obesity: magnetic resonance-based quantification of abdominal adipose tissue and liver fat in children. Rofo. 2012 Apr;184(4):324-32. doi: 10.1055/s-0031-1299094. Epub 2012 Feb 9. PMID 22322443
- [Result] Friebe D, Neef M, Kratzsch J, Erbs S, Dittrich K, Garten A, Petzold-Quinque S, Bluher S, Reinehr T, Stumvoll M, Bluher M, Kiess W, Korner A. Leucocytes are a major source of circulating nicotinamide phosphoribosyltransferase (NAMPT)/pre-B cell colony (PBEF)/visfatin linking obesity and inflammation in humans. Diabetologia. 2011 May;54(5):1200-11. doi: 10.1007/s00125-010-2042-z. Epub 2011 Feb 6. PMID 21298414
- [Result] Friebe D, Neef M, Erbs S, Dittrich K, Kratzsch J, Kovacs P, Bluher M, Kiess W, Korner A. Retinol binding protein 4 (RBP4) is primarily associated with adipose tissue mass in children. Int J Pediatr Obes. 2011 Jun;6(2-2):e345-52. doi: 10.3109/17477166.2010.491228. Epub 2010 Oct 15. PMID 20950077
- [Result] Korner A, Neef M, Friebe D, Erbs S, Kratzsch J, Dittrich K, Bluher S, Kapellen TM, Kovacs P, Stumvoll M, Bluher M, Kiess W. Vaspin is related to gender, puberty and deteriorating insulin sensitivity in children. Int J Obes (Lond). 2011 Apr;35(4):578-86. doi: 10.1038/ijo.2010.196. Epub 2010 Sep 21. PMID 20856257
- [Result] Ehehalt S, Wiegand S, Korner A, Schweizer R, Liesenkotter KP, Partsch CJ, Blumenstock G, Spielau U, Denzer C, Ranke MB, Neu A, Binder G, Wabitsch M, Kiess W, Reinehr T. Diabetes screening in overweight and obese children and adolescents: choosing the right test. Eur J Pediatr. 2017 Jan;176(1):89-97. doi: 10.1007/s00431-016-2807-6. Epub 2016 Nov 25. PMID 27888412
- [Result] Ehehalt S, Wiegand S, Korner A, Schweizer R, Liesenkotter KP, Partsch CJ, Blumenstock G, Spielau U, Denzer C, Ranke MB, Neu A, Binder G, Wabitsch M, Kiess W, Reinehr T. Low association between fasting and OGTT stimulated glucose levels with HbA1c in overweight children and adolescents. Pediatr Diabetes. 2017 Dec;18(8):734-741. doi: 10.1111/pedi.12461. Epub 2016 Nov 22. PMID 27873429
- [Result] Schreier M, Schwartze JT, Landgraf K, Scheuermann K, Erbs S, Herberth G, Pospisilik JA, Kratzsch J, Kiess W, Korner A. Osteopontin is BMI-independently Related to Early Endothelial Dysfunction in Children. J Clin Endocrinol Metab. 2016 Nov;101(11):4161-4169. doi: 10.1210/jc.2016-2238. Epub 2016 Aug 29. PMID 27571184
- [Result] Felix JF, Bradfield JP, Monnereau C, van der Valk RJ, Stergiakouli E, Chesi A, Gaillard R, Feenstra B, Thiering E, Kreiner-Moller E, Mahajan A, Pitkanen N, Joro R, Cavadino A, Huikari V, Franks S, Groen-Blokhuis MM, Cousminer DL, Marsh JA, Lehtimaki T, Curtin JA, Vioque J, Ahluwalia TS, Myhre R, Price TS, Vilor-Tejedor N, Yengo L, Grarup N, Ntalla I, Ang W, Atalay M, Bisgaard H, Blakemore AI, Bonnefond A, Carstensen L; Bone Mineral Density in Childhood Study (BMDCS); Early Genetics and Lifecourse Epidemiology (EAGLE) consortium; Eriksson J, Flexeder C, Franke L, Geller F, Geserick M, Hartikainen AL, Haworth CM, Hirschhorn JN, Hofman A, Holm JC, Horikoshi M, Hottenga JJ, Huang J, Kadarmideen HN, Kahonen M, Kiess W, Lakka HM, Lakka TA, Lewin AM, Liang L, Lyytikainen LP, Ma B, Magnus P, McCormack SE, McMahon G, Mentch FD, Middeldorp CM, Murray CS, Pahkala K, Pers TH, Pfaffle R, Postma DS, Power C, Simpson A, Sengpiel V, Tiesler CM, Torrent M, Uitterlinden AG, van Meurs JB, Vinding R, Waage J, Wardle J, Zeggini E, Zemel BS, Dedoussis GV, Pedersen O, Froguel P, Sunyer J, Plomin R, Jacobsson B, Hansen T, Gonzalez JR, Custovic A, Raitakari OT, Pennell CE, Widen E, Boomsma DI, Koppelman GH, Sebert S, Jarvelin MR, Hypponen E, McCarthy MI, Lindi V, Harri N, Korner A, Bonnelykke K, Heinrich J, Melbye M, Rivadeneira F, Hakonarson H, Ring SM, Smith GD, Sorensen TI, Timpson NJ, Grant SF, Jaddoe VW; Early Growth Genetics (EGG) Consortium; Bone Mineral Density in Childhood Study BMDCS. Genome-wide association analysis identifies three new susceptibility loci for childhood body mass index. Hum Mol Genet. 2016 Jan 15;25(2):389-403. doi: 10.1093/hmg/ddv472. Epub 2015 Nov 24. PMID 26604143
- [Result] Breitling C, Gross A, Buttner P, Weise S, Schleinitz D, Kiess W, Scholz M, Kovacs P, Korner A. Genetic Contribution of Variants near SORT1 and APOE on LDL Cholesterol Independent of Obesity in Children. PLoS One. 2015 Sep 16;10(9):e0138064. doi: 10.1371/journal.pone.0138064. eCollection 2015. PMID 26375028
- [Result] Qi Q, Downer MK, Kilpelainen TO, Taal HR, Barton SJ, Ntalla I, Standl M, Boraska V, Huikari V, Kiefte-de Jong JC, Korner A, Lakka TA, Liu G, Magnusson J, Okuda M, Raitakari O, Richmond R, Scott RA, Bailey ME, Scheuermann K, Holloway JW, Inskip H, Isasi CR, Mossavar-Rahmani Y, Jaddoe VW, Laitinen J, Lindi V, Melen E, Pitsiladis Y, Pitkanen N, Snieder H, Heinrich J, Timpson NJ, Wang T, Yuji H, Zeggini E, Dedoussis GV, Kaplan RC, Wylie-Rosett J, Loos RJ, Hu FB, Qi L. Dietary Intake, FTO Genetic Variants, and Adiposity: A Combined Analysis of Over 16,000 Children and Adolescents. Diabetes. 2015 Jul;64(7):2467-76. doi: 10.2337/db14-1629. Epub 2015 Feb 26. PMID 25720386
- [Result] Loffler D, Muller U, Scheuermann K, Friebe D, Gesing J, Bielitz J, Erbs S, Landgraf K, Wagner IV, Kiess W, Korner A. Serum irisin levels are regulated by acute strenuous exercise. J Clin Endocrinol Metab. 2015 Apr;100(4):1289-99. doi: 10.1210/jc.2014-2932. Epub 2015 Jan 27. PMID 25625801
- [Result] Mangner N, Scheuermann K, Winzer E, Wagner I, Hoellriegel R, Sandri M, Zimmer M, Mende M, Linke A, Kiess W, Schuler G, Korner A, Erbs S. Childhood obesity: impact on cardiac geometry and function. JACC Cardiovasc Imaging. 2014 Dec;7(12):1198-205. doi: 10.1016/j.jcmg.2014.08.006. Epub 2014 Oct 8. PMID 25306542
- [Result] Korner A, Wiegand S, Hungele A, Tuschy S, Otto KP, l'Allemand-Jander D, Widhalm K, Kiess W, Holl RW; APV initiative; German Competence Net Obesity. Longitudinal multicenter analysis on the course of glucose metabolism in obese children. Int J Obes (Lond). 2013 Jul;37(7):931-6. doi: 10.1038/ijo.2012.163. Epub 2012 Oct 2. PMID 23032406
- [Result] Ichimura A, Hirasawa A, Poulain-Godefroy O, Bonnefond A, Hara T, Yengo L, Kimura I, Leloire A, Liu N, Iida K, Choquet H, Besnard P, Lecoeur C, Vivequin S, Ayukawa K, Takeuchi M, Ozawa K, Tauber M, Maffeis C, Morandi A, Buzzetti R, Elliott P, Pouta A, Jarvelin MR, Korner A, Kiess W, Pigeyre M, Caiazzo R, Van Hul W, Van Gaal L, Horber F, Balkau B, Levy-Marchal C, Rouskas K, Kouvatsi A, Hebebrand J, Hinney A, Scherag A, Pattou F, Meyre D, Koshimizu TA, Wolowczuk I, Tsujimoto G, Froguel P. Dysfunction of lipid sensor GPR120 leads to obesity in both mouse and human. Nature. 2012 Feb 19;483(7389):350-4. doi: 10.1038/nature10798. PMID 22343897
- [Derived] Kempf E, Landgraf K, Vogel T, Spielau U, Stein R, Raschpichler M, Kratzsch J, Kiess W, Stanik J, Korner A. Associations of GHR, IGF-1 and IGFBP-3 expression in adipose tissue cells with obesity-related alterations in corresponding circulating levels and adipose tissue function in children. Adipocyte. 2022 Dec;11(1):630-642. doi: 10.1080/21623945.2022.2148886. PMID 36384443
- See also: Sonderforschungsbereich (SFB) Leipzig — https://www.sfb1052.de/
- See also: Link to Prof. Dr. med. Antje Körner's research group: "Childhood obesity" — http://kik.uniklinikum-leipzig.de/kikcms.site,postext,childhood-obesity-antje-koerner,a_id,1062.html
- See also: University Children's Hospital Leipzig (Germany) — http://kik.uniklinikum-leipzig.de/